CLINICAL TRIAL: NCT06247761
Title: StASSH TRAUMA - St Andrew's Study for Sutures in Trauma Hand Surgery Non Absorbable vs Absorbable Sutures in Trauma Hand Surgery- Does Choice of Suture Material Impact Wound Healing, Complication Rates or Patient Symptoms?
Brief Title: STASSH - TRAUMA - Absorbable vs Non-Absorbable Sutures in Trauma Hand Surgery
Acronym: STASSH-TRAUMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 328761
Record Dates: First submitted 2024-01-15; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Suture, Complication; Hand Infection; Skin Infection; Scar; Symptoms and Signs
Keywords: hand surgery; hand infection; complications; suture material; scar appearance
MeSH Terms: conditions — Cellulitis; Cicatrix; Signs and Symptoms

STUDY DESIGN:
Intervention Model Description: Single centre, parallel, two group, randomised control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vicryl rapide suture for Skin closure (Active Comparator): Skin closure at end of hand trauma surgery
  Interventions: Device: Skin closure at end of hand surgery
- Nylon suture for Skin closure (Active Comparator): Skin closure at end of hand trauma surgery
  Interventions: Device: Skin closure at end of hand surgery

INTERVENTIONS:
Device: Skin closure at end of hand surgery — skin closure with vicryl rapide suture

SUMMARY:
An RCT will be set up to compare outcomes between two groups of hand surgery patients. These are:

• Emergency hand surgery patients - randomized to either absorbable or non-absorbable suture.

The primary outcomes investigated will be:

• Infection occurrence

The secondary outcomes will be:

* Scar appearance at 1 week and 6-8 weeks (assessed from photographs and scar scoring scale)
* Wound inflammation as a percentage of wound length at day 7 post surgery.
* Patient symptoms at 1 week (assessed from patient questionnaire)
* Patient symptoms at 6-8 weeks (assessed from patient questionnaire)
* QDASH Score at 1 week (assessed from patient questionnaire)
* QDASH score at 6-8 weeks (assessed from patient questionnaire)
* Occurrence of other complications (assessed from the above photographs, the above questionnaires and from nurse and doctor led reports of wound breakdown and other complications)

DETAILED DESCRIPTION:
SUMMARY OF TRIAL DESIGN

This is a single-center, single-blinded, RCT with a parallel-group design to compare two groups of hand surgery patients.

TRIAL SETTING

The RCT will be a single- blinded single centre trial run at St. Andrew's Centre for Plastic and Reconstructive Surgery, Broomfield Hospital (part of MSEFT). St. Andrew's Centre is one of the busiest centres in the UK and plastic and reconstructive surgeons with many thousands of hand surgeries taking place every year.

Recruitment and Invitation

The Patient information sheet (PIS) will be provided to the patients that meet the criteria. If the patient declines, then it will be made clear that this will not affect their surgical or wound care.

The patients will have 48 hours minimum to read the PIS and to discuss and ask questions from our research team and the usual care team such as trauma clinic nurses, the research fellows, and consultants.

All patients will be asked on the day of surgery if they are happy to participate in the trial. If they agree to be in the trial, they will sign a consent form before the operation on the pre-operative ward.

If patients have concerns or require more information about the study, there will be provision for them to ask these questions in advance of the surgery day. The usual practice is to ask patients if they have any questions after each consultation to avoid information overload, unanswered questions, and anxiety. There will be no payments made to the participants to take part in this trial.

Images

Imaging (photographs) of the wounds are an integral part of this study. This will include a picture at 1 week post operation, and one picture 6-8 weeks post operation.

The images will be taken on a single digital camera. All photographs will be taken in the same clinic room in the dressing clinic, with the same lighting for each of the patients.

All images will be transferred to a password protected NHS Desktop folder at the end of each clinic day, and then deleted from the camera.

The images will then be saved on trust computers, in a trial specific password protected folder under the participants study ID and visit number (i.e. STASSH TRAUMA xxx - week 1).

The anonymised images of the wounds/scars may form part of the presentations, thesis and educational activities resulting from this project. A specific consent point has been included in the ICF to cover this research activity.

Patients involved in the trial may have health conditions that impact the healing of their wound, their scar appearance, and their symptoms.

The conditions known to impact wound healing are as follows:

* Diabetes
* Rheumatoid arthritis
* Ehlers-Danlos syndrome/connective tissue disorders
* Dermatological skin conditions effecting the hand e.g. eczema
* Patients on anticoagulant medication
* Patients taking immunosuppressant medication

All of the patient data will undergo stratification that will allow for a fair analysis to take place, which accounts for the higher risk of wound complications. Multivariate regression analysis will be undertaken in order to draw appropriate conclusions from the data which is collected.

Randomisation

On the morning of day of surgery randomisation will be carried out by the trauma clinic nurses/lead investigator. A simple sealed envelope randomisation process will be used.

There will be 480 envelopes in total. This ensures sufficient power for the study (400 minimum as per the reported 5% risk of infection from hand surgery), and takes into account potential withdrawals and lost to follow-up of 80/480 patients i.e. 40/240 from each of the two groups.

240 of these envelopes will be filled with a piece of paper marked with vicryl rapide suture, and 240 will be filled with a piece of paper marked nylon suture.

Which envelope is filled with which suture material type will be decided by a random number generator which will generate a number from 1-480, and each envelope will therefore be sequentially filled.

The trauma clinic nurse will have a supply of 480 sealed envelopes marked 'STASSH TRAUMA - randomisation number xxx' on the outside. These envelopes will be sequentially chosen in order to randomise participants to either the absorbable or non-absorbable group. This process will continue until 480 patients have been recruited into the study.

It is acknowledged that there may be some similarity between study ID and randomisation number therefore additional care will be taken by the research teams to record this data timely and accurately in the participants case report forms (CRFs).

For both groups, the patient will be blinded to the suture choice, and the operating team will be provided with the suture according to the group that the patient has been randomised to. As a result, the operating team will also be aware of the suture material being used.

The patient will be unblinded to suture allocation at day 7, when the non-absorbable group patients will require stitch removal. They will be required to complete the first part of the non-validated questionnaire, as well as the DASH questionnaire, BEFORE removal of their dressing. This is to ensure their reported symptoms are not biased by the appearance of the wound, or awareness of the suture type.

Blinding

Single blinding will be maintained by the patient's wound being covered with a dressing and bandage for the first week post operatively.

All theatre and clinic staff will be aware of which group the patient has been randomised to on the day of surgery. The sealed envelope will accompany the patient's notes into theatre and identify the suture material to be used for skin closure.

The type of suture material used will not be revealed to the patient (either vocally or in writing, before, during or after the surgery) but will be written in the operation note.

Data will be collected by staff in the dressing clinic, who are different to staff in the trauma clinic/hand surgery theatres. This will occur at 7 days and 42-56 days post operatively in dressing clinic and outpatient clinic respectively.

Patients will complete the first two questions in the non-validated questionnaire before removal of dressings. They will complete questions 3 and 4 of the non-validated questionnaire after removal of the dressing +/- stitch removal if indicated.

Patients will also be required to complete the DASH questionnaire before removal of the dressing takes place. This is essential to ensure that symptoms reported are not influenced by the patient or staff seeing the stitch material or appearance of the wound.

Unblinding

Although it is unlikely to be required over a short 7 day period, unblinding can be simply done by review of the participants medical or theatre notes or by unbandaging the participants hand where the choice of suture used would be obvious to clinical staff.

Any early unblinding will be recorded as a protocol deviation and would not be considered a withdrawal unless the participant expressly voices their desire to withdraw from the study.

Data Collection

Data will be collected throughout the surgery and during follow up periods. Project data collection will be managed by the research team and CI will oversee recruitment and collection of data. The CI will be responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported.

A folder will be kept in the dressing clinic and outpatient clinic areas. All completed patient questionnaires will be kept in this folder. The completed questionnaires will be collected from the folder at the end of the day and kept securely and onsite.

All data will be in anonymised form; patients will be identifiable only by study number and this will be sequentially allocated to patient at time of consent to participation on clinic day.

Surgical Procedure

All patients will undergo a hand surgery procedure. For the trauma cohort this will include tendon repairs, and open fractures. The only element of the surgery which will be affected by this study will be the skin closure at the very end of the surgery before dressings are applied. No study to date, has studied the effect of the structures impacted during hand surgery, on the wound healing process.

As mentioned before, there have been studies on carpal tunnel release surgery, and whether absorbable or non-absorbable sutures are superior. However there are significant limitations to this. Carpal tunnel surgery does not involve any tendons, blood vessels, nerves or ligaments. It is a 5-10 minute operation. Nobody to date has studied the effect of damaged tendons, nerves, blood vessels and ligaments on the skin healing process, and in particular if the choice of suture has an impact on wound healing in these cohorts.

The investigators are therefore adding first of its kind knowledge to the surgical literature, and will genuinely be able to inform guidance for trauma hand surgery. Any operating surgeon will be able to close the skin at the end of surgery, hence surgical acumen and seniority of the surgeon are not felt to be a factor in this study.

Post- Operative follow up face to face - day 7 and day 42-56 and end of study

Patients will be seen in dressing clinic at day 7 for photos, and for both the QDASH and non validated questionnaires to be filled. At day 7, the DASH questionnaire and the first part of the non-validated questionnaire must be completed before the dressings are removed and the patient is unblinded.

At day 42-56, the patient will be aware of the suture material already so any dressings can be removed before any questionnaires are completed.

Once the patient has completed the questionnaires, and has pictures of the wound taken, this defines the end of the study period for the patient.

STATISTICS

The power analysis for this study has been based on analysis by medical Statistician Dr Jufen Zhang of Anglia Ruskin Medical School. The primary outcome measure is wound infection. The sample size calculation is based on a 5% infection rate following hand surgery,

There are 480 (240 for each group) patients available in the study to compare differences between 2 groups.

The baseline continuous data will be summarised by the mean (standard deviation) or the median (25th - 75th percentile) depending on the distribution of data; categorical data by n (%). The difference between the two groups will be examined based on an intention-to-treat (ITT) principle.

The independent t-test or Mann-Whitey U test (depending on the distribution of the data) will be conducted to test if there is a difference in primary outcome variable between the two groups. The mean difference with 95% confidence intervals will be reported. A sensitivity analysis will be conducted to assess the robustness of the primary analysis to missing data.

Logistic regression models will be used to identify determinants for wound inflammation, complications, QDASH score and symptoms score. The study has more than 95% power to detect a "medium" effect size of 0.25 (Cohen, 1969) using one-way ANOVA with a significant level of 5%. Stata statistical computer package will be used to analyse the data.

Our primary outcome measure is infection rates, with other outcome measures being; wound inflammation as a proportion of wound length, scar appearance/score, QDASH score and patient symptoms.

No study to date has studied inflammation as a proportion of wound length following hand surgery. This is despite wound inflammation being an accurate predictor of pain from the wound, as well as accurate predictor of developing an infection. As such, it is not possible to perform a power calculation due to the paucity of the literature in this area.

For every patient, each of the outcomes the investigators are analysing will have a differential impact on their overall satisfaction with the surgery and the wound itself.

For some patients, wound appearance will be paramount. For others, the function of their hand (which the investigators will determine through the DASH and non validated questionnaires) is the most important factor, and for some the symptoms from the wound will have the biggest impact.

All of the primary and secondary outcome measures will be measured and analysed between the two groups, and will be appropriately stratified with the patients past medical conditions, use of post operative antibiotics, and the damaged structures in the surgery. Multivariate regression will be performed to account for any potential confounders and ensure a reliable analysis is performed.

This will ensure a fair comparison, and would be fairly and openly presented in any subsequent presentations or publications. It would be incorrect, to weigh one of the outcome measures more than the others, because every individual patient and surgeon values each of the outcomes differently.

PLANNED RECRUITMENT RATE

The aim will be to recruit 25 patients a week in one site i.e. St. Andrew's Centre for Plastic Surgery, MSEFT. This assumes a 20-30% recruitment rate (there are approximately 15 trauma operations occurring daily at MSEFT). Therefore, based on a sample size of 480 and 25 recruits per week, the recruitment period will be approximately 18-20 weeks.

WITHDRAWAL CRITERIA

The participant may withdraw their consent to continue in the study. If they withdraw their consent prior to treatment no further research activity will take place.

If the participant withdraws after the operation no further research activity will be undertaken and the participant will be followed-up according to standard care.

All data obtained prior to withdrawal will be retained as part of the study.

TRIAL MEDICATION

The sutures being used: polyglactin 910 (vicryl rapide), and ethilon (nylon), are already in widespread use across the NHS for a wide variety of surgeries. They are approved by the European Drug and Medicine authority.

Product Characteristics

VICRYL RAPIDE Suture, composed of 90% glycolide and 10% L-lactide copolymer, is a synthetic absorbable suture intended to model the performance of collagen (surgical gut) suture with less tissue reaction. It is indicated for use only in superficial soft tissue approximation of the skin and mucosa, with wound support of 7-10 days.

Vicryl sutures are among the preferred sutures of clinicians due to the low antigenicity, and sparse inflammatory infiltrates. Vicryl suture hypersensitivity is very rare. However, cases of suture allergies have been reported as pruritus, oedema, pain, and seroma formation. At the moment, no standardized method to test this reaction has been reported, and the rates of these complications is not reported in the literature. Hence the investigators have pioneered the measurement of inflammation as a proportion of wound length to measure this complication.

ETHILON Suture is a nonabsorbable, sterile surgical monofilament suture composed of the long-chain aliphatic polymers Nylon 6 and Nylon 6,6. ETHILON Suture is dyed black or green to enhance visibility in tissue. ETHILON Suture is indicated for use in general soft tissue approximation and/or ligation, including use in cardiovascular, ophthalmic, and neurological procedures. Only one incidence of adverse effects from nylon suture has rarely been reported in the literature, with the patient having erythema and pain until sutures were removed.

Product storage and supply

All sutures are stored in theatre and are kept in sterile packets. They are stored at room temperature.

They are simply opened onto a sterile trolley for the scrub nurse to load and give to the operating surgeon when the time for skin closure comes.

Products will be taken from standard hospital stocks, and will not add to theatre costs.

ELIGIBILITY:
Inclusion Criteria:

Adult emergency hand surgery patients (age 18-100) with suspected bone/tendon/nerve/blood vessel injury or high risk of infection e.g. bites

Exclusion Criteria:

* Patients who are unable to consent or do not consent
* Patients below the age of 18
* Patients with a known allergy to vicryl rapide (polyglactin 910) or nylon (ethilon) suture.
* Any patient whose hand surgery requires a skin graft.
* Any patient operated on as an immediate emergency e.g. amputation, revascularisation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-01-29 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Infection rate % | 6-8 weeks
  Infection rate %

SECONDARY OUTCOMES:
Wound inflammation | 1 week
  Measurement of erythema as a proportion of wound length using medical photography (unit is %, will be performed using photographic analysis and pixel counting software)
Scar appearance at 1 week | 1 week
  Scar appearance measured on Stony Brook Scar scale. 0 is worst score, 5 is best score.
Patient symptoms at 1 week | 1 week
  Non validated questionnaire. 4 item questionnaire, measured on scale of (3 is worst score, 15 is best score possible).
Patient symptoms at 6-8 weeks | 6-8 weeks
  Non validated questionnaire. 4 item questionnaire, measured on scale of (3 is worst score, 15 is best score possible).
Hand function at 1 week | 1 week
  QDASH (Quick disabilities of the Arm Shoulder and Hand) questionnaire (0 is best score, 10 is worst possible score)
Hand function at 6-8 weeks | 6-8 weeks
  QDASH (Quick disabilities of the Arm Shoulder and Hand) questionnaire (0 is best score, 10 is worst possible score)
Occurrence of any other complications | 6-8 weeks
  Reported complications during the duration of the trial participant inclusion in the study
Scar appearance at 6-8 weeks | 6-8 week
  Scar appearance measured on Stony Brook Scar scale. 0 is worst score, 5 is best score.

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD